CLINICAL TRIAL: NCT07348354
Title: Standardization and Application of Pure Platelet-Rich Plasma in Improving Sperm Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025.681
Record Dates: First submitted 2025-12-02; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This study will validate the standardized double-spin P-PRP protocol and evaluate its effect on sperm motility and DNA fragmentation after semen co-culture. It aims to enhance sperm quality while ensuring reproducibility and accessibility in clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-PRP group (Experimental): Sperm after washing without co-culture
  Interventions: Other: Standard culture
- PRP group (Experimental): Sperm after washing with PRP co-culture
  Interventions: Other: PRP culture

INTERVENTIONS:
Other: Standard culture — Only sperm culture
  Arms: Non-PRP group
Other: PRP culture — PRP 2-5% will be co-culture with sperm
  Arms: PRP group

SUMMARY:
Phase 1: Standardize and validate pure platelet-rich plasma (P-PRP) protocol

Aims:

To validate a standardized double-spin protocol for preparing pure platelet-rich plasma (P-PRP) in an IVF laboratory setting by assessing its platelet yield, purity, and reproducibility.

Outcomes

Primary outcome Platelet concentration in PRP Absolute platelet count in P-PRP and fold-increase compared to whole blood Secondary outcome Platelet recovery (%): (Platelet count in P-PRP × P-PRP volume) / (Whole blood platelet count × blood volume) × 100 Purity: White blood cell (WBC) concentration in P-PRP Growth factors :e.g.. VEGF, PDGF-AB, TGF-β, IGF-1… concentrations in plasma of PPP and P-PRP preparation Reproducibility Metrics: Coefficient of variation (CV%), intraclass correlation coefficient (ICC), and Bland-Altman limits of agreement for technical and biological duplicates.

Phase 2: Examine the effect of pure platelet-rich plasma (P-PRP) on sperm parameters Hypotheses and objectives Hypotheses The investigator hypothesizes that co-culture of semen with pure platelet-rich plasma (P-PRP) enhances sperm quality by increasing motility compared to standard culture medium without P-PRP (control group).

Primary outcome

- To compare total sperm motility after 24 hours of co-culture between semen samples co-cultured with P-PRP versus a control group (without P-PRP).

Secondary outcome

* To compare sperm parameters after other timepoints of co-culture between semen samples co-cultured with P-PRP versus a control group (without P-PRP).
* To compare the morphology and DNA Fragmentation Index (DFI) in semen samples after 24-hour co-culture with P-PRP versus control.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteer aged 18-45 years, willing to donate their blood
* Adequate sperm samples (raw sample TMS > 5 x 106)
* BMI <30 kg/m2

Exclusion Criteria:

* Concurrent administration of other agents such as prednisolone, intravenous immunoglobulin, or G-CSF
* Drug addiction
* Underlying uncontrolled genital infections, diabetes or hypertension, chromosomal or uterine abnormalities, genetic, hematologic, immunological, or endocrine disorders
* Chronic disease, systemic disease, or cancers
* Blood diseases (sepsis, thrombocytopenia)
* Do not agree to donate blood
* Use of supplements containing antioxidants within the past 3 months
* Administration of anticoagulants or NSAIDs at least 7 days before P-PRP infuse
* Haemoglobin < 11g/dL, platelet count < 150000 mm3

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-06-18 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
Phase I: Platelet concentration in PRP | Baseline
  Absolute platelet count in P-PRP
Phase II: total sperm motility | Up to 24 hours
  total sperm motility after 24 hours of co-culture between semen samples co-cultured with P-PRP versus a control group (without P-PRP).

SECONDARY OUTCOMES:
Phase I: Platelet recovery (%) | Baseline
  Platelet recovery (%)=(Platelet count in P-PRP × P-PRP volume) / (Whole blood platelet count × blood volume) × 100 in PRP
VEGF | Up to 8 weeks
  Growth factors VEGF concentration
TGF-β | Up to 8 weeks
  Growth factors PDGF-A concentration
IGF-1 | Up to 8 weeks
  Growth factors IGF-1concentration
Sperm progressive motility | Up to 24 hours
  Sperm progressive motility
Sperm non-progressive motility | Up to 24 hours
  Sperm non-progressive motility
Sperm immotility | Up to 24 hours
  Sperm immotility

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Chung Pui Wah Jacqueline, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No